CLINICAL TRIAL: NCT02024412
Title: The Safety and Effect of Monosialotetrahexosylganglioside Sodium Injection for Prevention Neurotoxicity of mFOLFOX6 as First-line Chemotherapy for Advanced Colorectal Cancer
Brief Title: Monosialotetrahexosylganglioside Sodium Injection for Prevention Neurotoxicity of mFOLFOX 6 in mCRC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20131123; E2013109A (Other: TianjinCIH)
Record Dates: First submitted 2013-11-24; First posted 2013-12-31 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Colorectal Cancer
Keywords: metastatic colorectal cancer; neurotoxicity; mFOLFOX6; monosialotetrahexosylganglioside Sodium Injection
MeSH Terms: conditions — Colorectal Neoplasms; Neurotoxicity Syndromes | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- monosialotetrahexosylganglioside Sodium (Experimental): arm A: monosialotetrahexosylganglioside Sodium Injection, 40mg,one hour before chemotherapy(mFOLFOX6), every two weeks until tumor progress or patients become intolerant
  Interventions: Drug: monosialotetrahexosylganglioside Sodium
- placebo (Placebo Comparator): arm B: equal saline as placebo ,one hour before chemotherapy(mFOLFOX6) every two weeks until tumor progress or intolerant
  Interventions: Other: placebo

INTERVENTIONS:
Drug: monosialotetrahexosylganglioside Sodium — it is a component extract from pig's brain,shenjie is the brand name
  Other Names: shenjie
  Arms: monosialotetrahexosylganglioside Sodium
Other: placebo — saline of the same appearance as monosialotetrahexosylganglioside Sodium
  Other Names: saline
  Arms: placebo

SUMMARY:
The morbidity of colorectal cancer(CRC) is 10%～15% in China.mFolfox6 has become one of the standard regimes for metastatic colorectal cancer (mCRC). Neutropenia and oxaliplatin-induced neurotoxicity are the most common adverse effects which even result in discontinue of chemotherapy, especially for patients suffered from heavily acute neurotoxicity. Monosialotetrahexosylganglioside is a component of membrane of nerve cells. Previous phase II clinical trial showed, it can reduce oxaliplatin-induced neurotoxicity(OIN). But it did not certificated by phase III trial. Investigators designed the phase III trial to investigate the effect and safety of monosialotetrahexosylganglioside Sodium Injection for prevention OIN at colorectal cancer.

DETAILED DESCRIPTION:
it is a placebo controlled phase III trial. investigators plan to enroll 240 patients with 1:1 to A arm and B arm

ELIGIBILITY:
Inclusion Criteria:

1. Patients shall have normal organic function such as liver function, Cardiac function and renal function;
2. age >18 years old;
3. diagnosis mCRC with histology;
4. Did not received first-line chemotherapy
5. Karnofsky Performance scores >70 scores
6. should have target lesions or non-target lesions
7. For patients received oxaliplatin before, the residual neurotoxicity should less than grade 2
8. For diabetes without neuropathy, blood glucose before meal should less than 8mmol/L and HBA1C<7.0%
9. Patients should be expected to live no shorter than 3 months

Exclusion Criteria:

1. patients who is receiving chemotherapy;
2. WBC<4.0×109/L，ANC<1.5×109/L,PLT<100×109/L，Hb<90g/L,TBIL>1.5Limitation;BUN）>1.5Limitation；Cr）>1.5Limitation；ALT or AST>2.5Limitation（without liver metastasis）；ALT or AST）>5Limitation（with liver metastasis）;
3. heart dysfunction;
4. brain metastasis;
5. peripheral nervous system or central nervous system abnormal including diabetes mellitus patients with neuropathy;
6. patients who received Glutathione, acetylcysteine, calcium / magnesium, amifostine, carbamazepine, B vitamins, vitamin E within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of neurotoxicity including acute neurotoxicity and accumulating neurotoxicity | From the first day of chemotherapy to 12 months after study or until one week before the patients receive second-line chemotherapy
  Acute neurotoxicity will be assessed the first day of oxaliplatin at every cycle given;accumulating neurotoxicity will be assessed every two weeks from the second day of first cycle until the patients out of the study. The accumulating neurotoxicity will be assessed every four weeks for 12 months or one week before second-line chemotherapy

SECONDARY OUTCOMES:
Objective response rate | Eevery 6 weeks, up to 24 months
  Investigators assess the effect every six weeks and objective response is recorded as complete response,partial response or stable disease according to Recist 1.1
Progress Free Survival | investigators assess the effect of chemotherapy every 6 weeks ,up to 24 months
  From date of randomization until the date of first documented progression
overall Survival | From date of randomization until the date of death from any cause, assessed up to 100 months
  the patients will be followed one month after progression ,then every 3 months,up to 100 months
quality of life | evaluate 1 week before chemotherapy and every 6 weeks of study. And evaluate within 4 weeks after the patients out of the study
  we use sf-36 to evaluated the quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ba, MD.PHD, Study Director — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China